CLINICAL TRIAL: NCT06659094
Title: Step Down From Maximal Support: Efficacy of Stepped-care Internet-based Cognitive Behavior Therapy for Obsessive-compulsive Disorder
Brief Title: Reducing Maximal Support in OCD: Efficacy of Stepped-Care Online CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-TX-004
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Obsessive Compulsive Disorder; Reduced-intensity stepped-care Internet-based Cognitive Behavioral Therapy; Randomized Controlled Trial; Cost effectiveness; Clinical Predictor
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stepped-care Internet-based cognitive behavioral therapy(SC-ICBT) combined with medication (Experimental): Patients' OCD severity is initially assessed with the Yale-Brown Obsessive Compulsive Scale (YBOCS). After enrollment, patients receive health education, observe symptoms, learn ERP theory, and create exposure lists on a WeChat mini-program for pre-treatment. They perform daily 1-hour ERP exercises for a week, with online status collection by coordinators. After a week, patients receive twice-weekly online ERP guidance from therapists for two weeks.
  After two and four therapy sessions, YBOCS re-evaluations occur via Tencent Meeting. Based on scores, the next three weeks involve either self-guided ERP or a mix of self-guided and therapist-guided ERP. If patients show over a 25% reduction, therapist guidance is suspended, and they switch to self-guided ICBT for the final three weeks.
  Interventions: Other: stepped-care Internet-based cognitive behavioral therapy(SC-ICBT); Drug: conventional medical treatment (TAU)
- Cognitive Behavioral Group Therapy (CBGT) combined with medication (Active Comparator): OCD patients will be provided with therapist-guided offline Cognitive Behavioral Group Therapy while they will continue with the medications they already have.
  A nationally registered psychotherapist, who has undergone systematic professional training, is in charge of a homogeneous closed group and records the sessions live. The treatment takes place in the group psychotherapy room at the Shanghai Mental Health Center, with a group of 6 people, for 6 weeks, twice a week, each session lasting 2 hours. A senior domestic group cognitive therapist supervises the treatment.
  Interventions: Other: Cognitive Behavioral Group Therapy (CBGT); Drug: conventional medical treatment (TAU)

INTERVENTIONS:
Other: stepped-care Internet-based cognitive behavioral therapy(SC-ICBT) — Using a WeChat mini-program, we offer personalized OCD SC-ICBT remote services. Training is customized based on individual assessments, focusing on psychological education and homework to simulate CBT therapy. If a patient's YBOCS score drop from baseline isn't 25% after four therapist sessions (one week of theory, two sessions/week), they get three more weeks of online guidance.
  The program includes four structured lessons over six weeks:
  Lesson 1: Psychological Health Education on OCD and related disorders. Lesson 2: ERP theory, exposure item lists, and related info. Lesson 3: Daily ERP practice for about an hour, followed by two weeks of therapist guidance.
  Lesson 4: Retrospection and relapse prevention.
  Arms: stepped-care Internet-based cognitive behavioral therapy(SC-ICBT) combined with medication
Other: Cognitive Behavioral Group Therapy (CBGT) — The CBGT group will receive cognitive-behavioral group therapy for 6 weeks, twice a week, each session lasting 2 hours, at the Shanghai Mental Health Center. The CBGT program follows a structured process for treating OCD. During the prep phase, therapists assess patients for 50 minutes, collect data, and set CBGT groundwork. In Session 1, families join to understand CBGT, with goals reinforced and OCD education provided. Session 2 reviews homework and develops ERP strategies. Session 3 initiates ERP practice. Sessions 4-11 continue homework review and group ERP practice. The final session involves families in a review, discussing challenges, celebrating achievements, and focusing on relapse prevention.
  Arms: Cognitive Behavioral Group Therapy (CBGT) combined with medication
Drug: conventional medical treatment (TAU) — Drug therapy, managed by a deputy chief psychiatrist unaware of patient groupings, utilizes China Food and Drug Administration (CFDA)-approved SSRIs for OCD. These include fluoxetine, paroxetine, sertraline, fluvoxamine, and others, with tricyclic drugs like clomipramine and SNRIs such as venlafaxine. The maximum dosage adheres to the instructions. Benzodiazepines may assist with sleep, but usage is capped at two weeks; no other psychotropics are co-administered. Common side effects comprise dry mouth, constipation, nausea, indigestion, dizziness, fatigue, and sweating. The maximum dosage shall not exceed the maximum dosage prescribed in the instruction manual.

SUMMARY:
This study is conducted to explore the efficacy and cost-effectiveness of stepped-care internet-based cognitive behavior therapy (sc-ICBT) with reduced support compared to cognitive-behavioral group therapy(CBGT), to identify the optimal transition points for shorter effective stepped treatments, to find clinical indicators that can predict the effectiveness of CBT interventions, and to investigate predictive outcomes.

The main questions the investigators aim to answer are:

1. Is the reduction in YBOCS scores following stepped-care Internet-based cognitive-behavioral therapy (SC-ICBT) with reduced support non-inferior to that observed in traditional cognitive-behavioral group therapy (CBGT)?
2. Does SC-ICBT for obsessive-compulsive disorder offer better health economic benefits compared to CBGT?
3. What is the optimal time point for transitioning to shorter effective stepped care, and what clinical indicators can predict the efficacy of CBT interventions post-treatment?

DETAILED DESCRIPTION:
SC-ICBT is a therapy combining therapist-guided and semi-self-directed ICBT, with treatment plans adjusted based on patient symptoms. While it aims to be minimally restrictive and low-cost, research shows that low-intensity treatment may miss the mark for patients with severe symptoms or low motivation. High dropout rates and safety concerns are also noted. To address this, the investigators propose starting with high-intensity one-on-one support, reassessing symptoms in the third week, and switching to low-intensity self-guided practice if improvement is seen, otherwise continuing high-intensity support.

In our study, the investigators will conduct a stepped-care Internet-based Cognitive Behavioral Therapy (ICBT) intervention trial with reduced support intensity: Following baseline symptom assessment (Week 0), participants will be allocated to either an online therapy group or an in-person group therapy group. Considering practicality, the study will employ a partially randomized allocation method: for participants who are convenient for both treatment modalities, the investigators will use random numbers to randomly assign them to either the online therapy group or the in-person group therapy group; if participants can only attend one of the treatment groups, the investigators will allocate them based on their preference. The group assignment will be blinded to the assessors. The study will feature two groups for a controlled trial: the experimental group, stepped-care ICBT combined with medication; the control group, cognitive-behavioral group therapy combined with medication. This study is conducted to explore the efficacy and cost-effectiveness of sc-ICBT with reduced support compared to CBGT in China.

The investigators plan to recruit 80 patients and assign them to the SC-ICBT group and the CBGT group for a 6-week intervention, with a follow-up period of 3 months post-intervention. During this period, the investigators will employ questionnaires, scales, functional magnetic resonance imaging (fMRI), and other experimental methods to assess participants' obsessive-compulsive symptoms and treatment outcomes. Concurrently, the investigators will collect data on patients' economic burden and self-reported health status to evaluate the cost effect of SC-ICBT.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged between 18 and 50 years, inclusive of both genders;
2. Presenting primarily with compulsive symptoms that meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Obsessive-Compulsive Disorder (OCD);
3. Yale-Brown Obsessive Compulsive Scale (YBOCS) scores ranging from 16 to 31, inclusive;
4. Have been on a stable regimen of standard anti-compulsive pharmacotherapy for a period of 8 weeks;
5. Possess a minimum educational level of junior high school;
6. Demonstrate adequate auditory and visual acuity to perform the assessments required by the study;
7. The participant and their legal guardian have comprehended the nature of the study and have provided informed consent;
8. Right-handedness (this criterion applies exclusively to participants undergoing magnetic resonance imaging).

Exclusion Criteria:

1. Satisfied with the diagnostic criteria for a mental disorder in DSM-V other than OCD.
2. Obsessive-compulsive symptoms were too severe to participate in the experiment.
3. High risk of suicide.
4. Severe central system or physical disease
5. Pregnant women or women that getting ready for being pregnant and lactating.
6. Other treatments being performed.
7. Uncooperative or unable to complete treatment
8. With metal implants in the body, such as pacemakers, intracranial silver clips, metal dentures, arterial stents, arterial clips, joint metal fixation, or other metal implants, etc. (this criterion is for fMRI subjects only)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change of Yale-Brown Obsessive-Compulsive Scale (YBOCS) | Change from Baseline at 6 weeks
  YBOCS is compiled by Goodman in the United States and contains 10 items to assess the severity of obsessive thoughts and compulsive behavior. The scoring method adopts a five-point scale of 0-4 points, and the total score range is 0-40 points, which has good reliability and validity. Scores below 16 are considered mild or subclinical, 16 to 23 points indicate moderate severity, 24 to 31 points indicate severe severity, and scores above 31 indicate extremely severe.

SECONDARY OUTCOMES:
Change of Florida Obsessive-Compulsive Inventory (FOCI) | Change from Baseline at 6 weeks
  FOCI, a self-rating scale, is used to assess the severity of obsessive-compulsive symptoms within one month, which contains 20 items. The first 15 items are evaluated the symptoms by yes and no, and the last 5 items are evaluated the severity of symptoms on 0-4 five-point scale. The Chinese version of the FOCI severity scale ≥8 is considered positive (i.e., indicative of obsessive-compulsive disorder).
Change of Self-rating Depression Scale (SDS) | Change from Baseline at 6 weeks
  The Self-Rating Depression Scale (SDS) was developed by William W. K. Zung from the Duke University School of Medicine in 1965 and is one of the most widely used self-assessment scales for depression. It is used to measure the severity of depressive states and their changes during treatment.
  According to the Chinese norm results, the cutoff value for the SDS standard score is 53 points, with 53-62 points indicating mild depression, 63-72 points indicating moderate depression, and above 73 points indicating severe depression. The normal upper limit for the SDS total raw score is 41 points, with lower scores indicating a better state. The standard score is the integer part obtained by multiplying the total raw score by 1.25. In China, a SDS standard score ≥50 is considered to have depressive symptoms.
Change of Self-rating Anxiety Scale (SAS) | Change from Baseline at 6 weeks
  The Self-rating Anxiety Scale (SAS) is very similar to the Self-rating Depression Scale (SDS) from the scale construction to the evaluation method. It is a very simple clinical tool to analyze the subjective anxiety symptoms of patients. It is suitable for adults with anxiety symptoms and has a wide range of application.According to the Chinese norm results, the cut-off value for SAS standard deviation is 50 points, with 50-59 points indicating mild anxiety, 60-69 points indicating moderate anxiety, and above 69 points indicating severe anxiety.
The University of Rhode Island Change Assessment | Change from Baseline at 6 weeks
  The University of Rhode Island Change Assessment (URICA) is a self-report measurement method developed by McConnaughy, DiClemente, Prochaska, and Velicer . The 24-item version consists of four dimensions: Precontemplation (Cronbach's α = 0.79), Contemplation (Cronbach's α = 0.84), Action (Cronbach's α = 0.84), and Maintenance (Cronbach's α = 0.82). URICA is commonly used to study motivation related to the treatment of behavioral health issues, and few studies have explored the specific relationship between the URICA scales and Cognitive Behavioral Therapy (CBT) for obsessive-compulsive disorder.For the general population, the following cut-off scores may be appropriate:
  8 or lower classified as People in Precontemplation 8-11 classified as People in Contemplation 11-14 classified as People in Preparation or Action For intensive service populations, it may be more appropriate to use only score in the range of 12-14 to classify those in preparation and action.

OTHER OUTCOMES:
Short-Form 6-Dimension Health Survey Version 2 (SF-6Dv2) | Change from Baseline at 6 weeks
  The full name of the self-completed Six-Dimension Health Survey Brief Form (SF-6Dv2) is "Short Form Six-Dimensions version 2". The SF-6Dv2 is an updated version of the widely used SF-36 Health Survey Questionnaire. It is a health utility measurement tool used to assess an individual's health-related quality of life (HRQoL) and convert it into health utility values, which can be used to calculate Quality Adjusted Life Years (QALYs). The SF-6Dv2 includes six dimensions: physical function, role limitation, social function, pain, mental health, and vitality.
Cost-effectiveness analysis | The cost from Baseline to Week 6
  The study designs a self-rated questionnaire about cost-effectiveness analyses, including both direct and indirect costs, and the patients themselves fill out the questionnaire based on the bill. The cost-effectiveness analysis method (CEA) is used to measure the spending of three groups. The results of the total cost divided by YBOCS total reduction scores can reflect the cost required to obtain each unit of curative effect.
Cost-utility analysis | The cost from Baseline to Week 6
  The cost-utility analysis method is used to measure the spending of improving patients' quality of life. The results of the total cost divided by SF-36 total improvement scores can reflect the cost required to obtain each unit of utility.
Dropout rate | From Baseline to Week 6
  Dropout rate is recorded to evaluate treatment acceptability.
Frequency of occurrence | From Baseline to Week 6
  Frequency of occurrence is recorded to evaluate treatment acceptability. The investigators use sign-in sheets to measure patients' attendance during the treatment.
Homework completion | From Baseline to Week 6
  Homework completion is recorded to evaluate treatment acceptability. The investigators use sign-in sheets to keep track of patients' homework completion.
Subjective satisfaction with treatment | From Baseline to Week 6
  Subjective satisfaction with treatment is recorded to evaluate treatment acceptability. The investigators use a self-rated question（"Overall, how satisfied are you with your current treatment?") to measure patients' subjective satisfaction. The rating was done on a 7-item scale ranging from "Extremely dissatisfied" to "Extremely satisfied".
Treatment safety | From Baseline to Week 6
  Adverse events (AEs) are the treatment safety indicators
Change of randomized dot motion(RDM) perceptual decision-making task | Change from Baseline at 6 weeks
  RDM is a classic perceptual decision-making paradigm where participants are required to report the overall direction of motion of 300 randomly moving white dots, with the total task duration being approximately 25 minutes. RDM is often used in conjunction with the drift diffusion model to study human decision-making processes and has been supported by a wealth of research evidence . Following the RDM decision, a confidence assessment phase is added, measuring participants' decision confidence through their subjective reports.
Change of the antisaccade task | Baseline and Week 6
  Anti-saccade task is a behavioral paradigm measuring response inhibition ability. Each trial started with a red or green central disc (1°diameter), lasting for 450/600/750/900ms. Participants were instructed to fixate on the central disc. The color (red vs. green) indicated whether the current trial was prosaccade or antisaccade, and the mapping between the color and the trial type was counterbalanced across participants. Then, together with the central disc, a white disc (1° diameter) was presented for 500ms at the left or right border of the grey rectangle. Participants were required to look at the white disc with their eyes given a prosaccade trial, and to look at the opposite location given an anti-saccade trial. Participants were instructed to respond as accurately and quickly as possible. A blank screen of 1500 ms was presented after the target. There were 40 trials in each condition. The total 80 trials were mixed and divided into 4 blocks of equal length.
Change of the task-state functional magnetic resonance imaging(fMRI) of the whole brain | Change from Baseline at 6 weeks
  The investigators use the randomized dot motion perceptual decision-making task as Neuroimaging Paradigm to observe the neurophysiological changes cauesd by step-ICBT in patients with OCD.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Fan, Doctor, Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China